CLINICAL TRIAL: NCT03641209
Title: Extremely Low Gestational Age Infants' Paracetamol Study: a Randomized Trial
Brief Title: Extremely Low Gestatonal Age Infants' Paracetamol Study
Acronym: Paras
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Outi Aikio (Other)
Responsible Party: Sponsor-Investigator, Outi Aikio, MD, PhD, Docent, Specialist in pediatrics and neonatology, University of Oulu
Organization: University of Oulu (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 39/2018
Record Dates: First submitted 2018-08-03; First posted 2018-08-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Prematurity; Extreme; Low Birthweight, Extremely (999 Grams or Less)
Keywords: acetaminophen; ductus arteriosus; NIRS; intravenous
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, one center trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo, 0.45 % saline, is similar to paracetamol, both being clear liquids, so the staff will remain unaware which drug the patient receives. The study drug will be kept and prepared away from the NICU, at the separate ward 55 office, in a locked cabinet. The study drug will be prepared by the research nurse, the pharmacist of the ward, or during nighttime, by a nurse who does not participate in the study patients' treatment in any way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol 10 mg/mL infusion solution, intravenous loading dose 20 mg/kg, followed by maintenance dose 7.5 mg/kg every 6 h up to 9 days
  Interventions: Drug: Paracetamol 10mg/mL infusion solution
- Placebo (Placebo Comparator): 0.45% sodium chloride (NaCl) solution, equal amounts in mL as would have been given the experimental drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Paracetamol 10mg/mL infusion solution — Intravenous paracetamol solution for infusion
  Other Names: acetaminophen; Paracetamol Fresenius Kabi 10 mg/mL infusion solution
  Arms: Paracetamol
Other: Placebo — Half physiological saline solution as the non-active placebo solution
  Other Names: Natriumklorid Braun 4,5mg/mL solution for infusion
  Arms: Placebo

SUMMARY:
In the present trial, early, intravenous paracetamol is compared to placebo in extremely premature or low birth weight infants in order to evaluate the effect on ductal closure.

DETAILED DESCRIPTION:
The purpose of this randomized, placebo-controlled, double-blind, phase 2, one center clinical trial is to study the efficacy and safety of early (< 96 h) intravenous paracetamol in prophylactic closure of ductus arteriosus in extremely premature (gestational age <28+0 wk, ELGA) or low birth weight (<1000 g, ELBW) infants. The infants born extremely preterm or low birth weight are a focus of the study, since a small phase 2 study on paracetamol failed to demonstrate contraction of ductus arteriosus.

In the investigator's previous cohort of ELGA/ELBW infants, the numbers of patients who needed any therapies for patent ductus arteriosus (PDA) were 29 (23%) in the paracetamol exposed group, and 90 (54%) in the control group. As demonstrated in a phase 2 study, the early paracetamol treatment induced the closure of ductus arteriosus: the mean (SD) ductal closure age was 177 (338) h in the whole paracetamol group. However, in the subgroup of ELGA infants born before 28 gestation weeks (n=14), the mean (SD) ductal closure ages in the paracetamol and placebo groups were 491 (504) h and 858 (719) h, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born before 28+0 gestation weeks and/or birth weight less than 1000g

Exclusion Criteria:

* Severe malformation or suspected chromosomal defect or other very severe life-threatening disease (e.g. very severe birth asphyxia or persistent pulmonary hypertension, etc.)

Max Age: 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Ductal closure | Neonatal intensive care unit (NICU) treatment period up to 13 weeks
  Postnatal age of the observed closure of ductus arteriosus

SECONDARY OUTCOMES:
Near-infrared spectroscopy values | Study drug period up to 10 days
  Near-infrared spectroscopy values
Paracetamol serum levels | Study drug period up to 10 days
  Paracetamol serum levels
Paracetamol side effects | Neonatal intensive care unit (NICU) treatment period up to 13 weeks
  Any observed or detected paracetamol side effects
PDA | Neonatal intensive care unit (NICU) treatment period up to 13 weeks
  Open ductus arteriosus without any traditional PDA therapies
PDA, treated | Neonatal intensive care unit (NICU) treatment period up to 13 weeks
  The need for PDA therapies (ibuprofen, paracetamol, ligation)
Ventilatory assist | Neonatal intensive care unit (NICU) treatment period up to 13 weeks
  The duration of any ventilation assist, days
Complications of prematurity | The first hospitalization period up to 19 weeks
  The long term complications of prematurity (moderate-to-severe bronchopulmonary dysplasia (BPD), intraventricular hemorrhage gr 2-4, moderate to severe necrotizing enterocolitis, retinopathy of prematurity (ROP) needing therapy)
Long term morbidity | The first hospitalization period up to 19 weeks
  Other long-term morbidity
Mortality | The first hospitalization period up to 19 weeks
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Outi Aikio, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Department of Pediatrics, Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juujarvi S, Saarela T, Hallman M, Aikio O. Intravenous paracetamol was associated with closure of the ductus arteriosus in extremely premature infants. Acta Paediatr. 2018 Apr;107(4):605-610. doi: 10.1111/apa.14137. Epub 2017 Nov 17. PMID 29105147
- [Background] Harkin P, Harma A, Aikio O, Valkama M, Leskinen M, Saarela T, Hallman M. Paracetamol Accelerates Closure of the Ductus Arteriosus after Premature Birth: A Randomized Trial. J Pediatr. 2016 Oct;177:72-77.e2. doi: 10.1016/j.jpeds.2016.04.066. Epub 2016 May 20. PMID 27215779
- [Background] Harma A, Aikio O, Hallman M, Saarela T. Intravenous Paracetamol Decreases Requirements of Morphine in Very Preterm Infants. J Pediatr. 2016 Jan;168:36-40. doi: 10.1016/j.jpeds.2015.08.003. Epub 2015 Aug 29. PMID 26323200
- [Background] Aikio O, Harkin P, Saarela T, Hallman M. Early paracetamol treatment associated with lowered risk of persistent ductus arteriosus in very preterm infants. J Matern Fetal Neonatal Med. 2014 Aug;27(12):1252-6. doi: 10.3109/14767058.2013.854327. Epub 2013 Oct 31. PMID 24111688

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03641209/Prot_SAP_000.pdf